CLINICAL TRIAL: NCT03341208
Title: Quantitative Assessment of Right Ventricular Strain Utilizing Cardiac Magnetic Resonance Imaging: Development of an Optimal Measure of Treatment Response Following Catheter-directed Interventions on Sub-massive Pulmonary Embolism.
Brief Title: Quantitative Assessment of RV Strain Using cMRI Following Catheter Intervention on PE
Acronym: RVEF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Charles Hennemeyer, Chief Vascular and Interventional Radiology, University of Arizona
Other Study IDs: UArizonaIR
Record Dates: First submitted 2017-11-07; First posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Right Ventricular Failure; Pulmonary Embolism
MeSH Terms: conditions — Heart Failure; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cardiac Magnetic Resonance Imaging — Cardiac MRI will be performed before and after subject has undergone catheter directed therapy

SUMMARY:
Acute pulmonary embolism (PE) is a condition in which the vessels carrying blood to the lungs become suddenly blocked, usually by a blood clot. There are a number of adverse consequences that result, with one of the most significant being strain on the right side of the heart (which must push blood through the blocked arteries to the lungs). Although this strain on the right heart is very important, current methods for measuring it are flawed. The standard practice is to obtain an echocardiogram (ultrasound of the heart), from which indirect measurements of the size of the heart are used to make inferences about right heart strain. This method can help guide management in some patients, but it in not a sensitive test and does not provide detailed information.

Patients with PE are treated with blood thinning medications. Some patients may be referred to the Interventional Radiology (IR) team for endovascular intervention, in which catheters are placed into the patient's vessels under radiologic guidance and advanced to the lungs to remove the clot entirely.

Cardiac magnetic resonance imaging (MRI) is a well-established imaging technique that produces highly detailed images of the heart's structure and function, with no risks to patients of ionizing radiation or intravenous contrast. Cardiac MRI is far superior to echocardiogram in evaluation of the right side of the heart, however it has not been widely used in the evaluation of patients with PE. We propose that by using a fast MRI protocol, we will be able to detect right heart strain with more accuracy than echocardiogram. Furthermore, we hypothesize that MRI images obtained before and after IR catheter-directed therapy will demonstrate the degree to which strain is relieved with this treatment. Finally, we believe that using MRI may help to guide management of patients with PE by detecting early or mild heart strain before it progresses.

In order to test these hypotheses, we plan to image PE patients who have been referred to the IR team with MRI. Patients recruited for this study will undergo two short MRI scans - one immediately before treatment, and one after completion of IR treatment (which lasts approximately 12-24 hours).

DETAILED DESCRIPTION:
Pulmonary embolism occurs when embolic material (usually clot in the venous system) travels to the heart and lodges in the pulmonary vasculature. This obstruction, if significant, can lead to pulmonary arterial hypertension, which places increased demand on the right ventricle (RV), which must pump against the blockage. This can manifest as right ventricular dysfunction (RVD), which is characterized by dilatation of the RV, wall motion abnormalities and other structural and functional changes. There is a significant body of data demonstrating that function of the RV is an important prognostic indicator in patients with acute PE. In these studies, RVD allowed identification of patients who, although clinically stable on presentation, were at risk for hemodynamic instability and high morbidity/mortality. As a result, many authors have suggested that RVD represents an important indication for more aggressive therapy in patients with submassive PE.

Currently, echocardiography is the most commonly used method for evaluating the RV in acute PE. However, obtaining quality imaging of the RV using echocardiography is technically difficult, and determining a reliable indicator of RV function has proved challenging. A number of markers of right ventricular function have been described, including size criteria, ejection fraction, wall motion, tricuspid regurgitation, paradoxical septal motion, and others. However, there is no general consensus on which methodology or measurements produce the most clinically meaningful data. The American Heart Association guidelines for submassive pulmonary embolism use the ratio of the right ventricle to left ventricle at end diastole (RV:LV ratio), which is defined as greater than 0.9 in patients with RVD. However, there is a large degree of heterogeneity in echocardiographic criteria for RVD used in the literature.

Additionally, the quantitative data provided by echocardiography is suspect, as they show only modest correlation with cardiac magnetic resonance imaging (cMRI) or computed tomography (CT) in evaluation of the RV. Even when specifically utilizing the American Society of Echocardiography guidelines, echocardiography proves to be significantly less accurate than cMRI for evaluation of the RV, especially in patients with a dilated ventricle.

Cardiac magnetic resonance imaging is considered the reference standard for accurate evaluation of ventricular structure and function. It has proven its accuracy, reliability, and prognostic value in the setting of other pathologies that result in RV dysfunction, such as pulmonary hypertension. However, to date, this modality has not been used to provide detailed information about the structure and function of the RV in patients with acute PE.

Recently, new therapies for acute PE have come into use that allow more precise treatment of the embolus itself through the use of endovascular catheters. These catheter-directed therapies (CDTs) deliver thrombolytic medication or other treatment strategies directly to the pulmonary circulation. There is a strong body of evidence supporting the use of these therapies, and some devices have been FDA-approved for this indication. Despite this, there is a lack of definitive markers for the patients who would benefit most from this therapy. Additionally, techniques currently used to attempt to quantify response to therapy (such as RV:LV ratio) are not ideal. There remains a need for a quantitative method for evaluating the structure and function of the RV in patients with acute PE in order to determine their risk for hemodynamic compromise, the need for CDT, and response after therapy is completed.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be patients who present to the emergency department or are inpatients in the hospital, who are found to have a diagnosis of acute pulmonary embolism (confirmed by computed tomography pulmonary angiography), and who have been referred to Interventional Radiology for evaluation for CDT. Patients appropriate for recruitment into this study will have large PEs involving lobar branches or more central segments of the pulmonary arteries.

Exclusion Criteria:

* Exclusion criteria will be limited to prisoners, pregnant women, patients for whom English or Spanish is not a first language, severe claustrophobia, and other routine contraindications for MRI. Patients with massive PE (resulting in hemodynamic instability) will not be appropriate participants for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 10 patients will be recruited for the study. Participants will be patients who present to the emergency department or are inpatients in the hospital, who are found to have a diagnosis of acute pulmonary embolism (confirmed by computed tomography pulmonary angiography), and who have been referred to Interventional Radiology for evaluation for CDT. Patients appropriate for recruitment into this study will have large PEs involving lobar branches or more central segments of the pulmonary arteries. However, patients with massive PE (resulting in hemodynamic instability) will not be appropriate participants for this study.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Measure RVEF prior to and after catheter directed therapy to remove pulmonary thromboembolus | 2 years
  Will predict severity of PE and identify patients that would most benefit from catheter therapy

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hennemeyer, MD, Principal Investigator — University of Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lualdi JC, Goldhaber SZ. Right ventricular dysfunction after acute pulmonary embolism: pathophysiologic factors, detection, and therapeutic implications. Am Heart J. 1995 Dec;130(6):1276-82. doi: 10.1016/0002-8703(95)90155-8. PMID 7484782
- [Background] Grifoni S, Olivotto I, Cecchini P, Pieralli F, Camaiti A, Santoro G, Conti A, Agnelli G, Berni G. Short-term clinical outcome of patients with acute pulmonary embolism, normal blood pressure, and echocardiographic right ventricular dysfunction. Circulation. 2000 Jun 20;101(24):2817-22. doi: 10.1161/01.cir.101.24.2817. PMID 10859287
- [Background] Fremont B, Pacouret G, Jacobi D, Puglisi R, Charbonnier B, de Labriolle A. Prognostic value of echocardiographic right/left ventricular end-diastolic diameter ratio in patients with acute pulmonary embolism: results from a monocenter registry of 1,416 patients. Chest. 2008 Feb;133(2):358-62. doi: 10.1378/chest.07-1231. Epub 2007 Oct 20. PMID 17951624
- [Background] Cho JH, Kutti Sridharan G, Kim SH, Kaw R, Abburi T, Irfan A, Kocheril AG. Right ventricular dysfunction as an echocardiographic prognostic factor in hemodynamically stable patients with acute pulmonary embolism: a meta-analysis. BMC Cardiovasc Disord. 2014 May 6;14:64. doi: 10.1186/1471-2261-14-64. PMID 24884693
- [Background] Jurcut R, Giusca S, La Gerche A, Vasile S, Ginghina C, Voigt JU. The echocardiographic assessment of the right ventricle: what to do in 2010? Eur J Echocardiogr. 2010 Mar;11(2):81-96. doi: 10.1093/ejechocard/jep234. Epub 2010 Feb 2. PMID 20124362
- [Background] Wake N, Kumamaru KK, George E, Bedayat A, Ghosh N, Gonzalez Quesada C, Rybicki FJ, Gerhard-Herman M. Computed tomography and echocardiography in patients with acute pulmonary embolism: part 1: correlation of findings of right ventricular enlargement. J Thorac Imaging. 2014 Jan;29(1):W1-6. doi: 10.1097/RTI.0000000000000047. PMID 24157621
- [Background] Jaff MR, McMurtry MS, Archer SL, Cushman M, Goldenberg N, Goldhaber SZ, Jenkins JS, Kline JA, Michaels AD, Thistlethwaite P, Vedantham S, White RJ, Zierler BK; American Heart Association Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation; American Heart Association Council on Peripheral Vascular Disease; American Heart Association Council on Arteriosclerosis, Thrombosis and Vascular Biology. Management of massive and submassive pulmonary embolism, iliofemoral deep vein thrombosis, and chronic thromboembolic pulmonary hypertension: a scientific statement from the American Heart Association. Circulation. 2011 Apr 26;123(16):1788-830. doi: 10.1161/CIR.0b013e318214914f. Epub 2011 Mar 21. PMID 21422387
- [Background] Pruszczyk P, Goliszek S, Lichodziejewska B, Kostrubiec M, Ciurzynski M, Kurnicka K, Dzikowska-Diduch O, Palczewski P, Wyzgal A. Prognostic value of echocardiography in normotensive patients with acute pulmonary embolism. JACC Cardiovasc Imaging. 2014 Jun;7(6):553-60. doi: 10.1016/j.jcmg.2013.11.004. Epub 2014 Jan 8. PMID 24412192
- [Background] Kjaergaard J, Petersen CL, Kjaer A, Schaadt BK, Oh JK, Hassager C. Evaluation of right ventricular volume and function by 2D and 3D echocardiography compared to MRI. Eur J Echocardiogr. 2006 Dec;7(6):430-8. doi: 10.1016/j.euje.2005.10.009. Epub 2005 Dec 9. PMID 16338173
- [Background] Lai WW, Gauvreau K, Rivera ES, Saleeb S, Powell AJ, Geva T. Accuracy of guideline recommendations for two-dimensional quantification of the right ventricle by echocardiography. Int J Cardiovasc Imaging. 2008 Oct;24(7):691-8. doi: 10.1007/s10554-008-9314-4. Epub 2008 Apr 28. PMID 18438737
- [Background] Mooij CF, de Wit CJ, Graham DA, Powell AJ, Geva T. Reproducibility of MRI measurements of right ventricular size and function in patients with normal and dilated ventricles. J Magn Reson Imaging. 2008 Jul;28(1):67-73. doi: 10.1002/jmri.21407. PMID 18581357
- [Background] van Wolferen SA, Marcus JT, Boonstra A, Marques KM, Bronzwaer JG, Spreeuwenberg MD, Postmus PE, Vonk-Noordegraaf A. Prognostic value of right ventricular mass, volume, and function in idiopathic pulmonary arterial hypertension. Eur Heart J. 2007 May;28(10):1250-7. doi: 10.1093/eurheartj/ehl477. Epub 2007 Jan 22. PMID 17242010
- [Background] Benza R, Biederman R, Murali S, Gupta H. Role of cardiac magnetic resonance imaging in the management of patients with pulmonary arterial hypertension. J Am Coll Cardiol. 2008 Nov 18;52(21):1683-92. doi: 10.1016/j.jacc.2008.08.033. PMID 19007687
- [Background] Alunni JP, Degano B, Arnaud C, Tetu L, Blot-Souletie N, Didier A, Otal P, Rousseau H, Chabbert V. Cardiac MRI in pulmonary artery hypertension: correlations between morphological and functional parameters and invasive measurements. Eur Radiol. 2010 May;20(5):1149-59. doi: 10.1007/s00330-009-1664-3. Epub 2010 Jan 22. PMID 20094890
- [Background] Sista AK, Kearon C. Catheter-Directed Thrombolysis for Pulmonary Embolism: Where Do We Stand? JACC Cardiovasc Interv. 2015 Aug 24;8(10):1393-1395. doi: 10.1016/j.jcin.2015.06.009. No abstract available. PMID 26315744
- [Background] Kucher N, Boekstegers P, Muller OJ, Kupatt C, Beyer-Westendorf J, Heitzer T, Tebbe U, Horstkotte J, Muller R, Blessing E, Greif M, Lange P, Hoffmann RT, Werth S, Barmeyer A, Hartel D, Grunwald H, Empen K, Baumgartner I. Randomized, controlled trial of ultrasound-assisted catheter-directed thrombolysis for acute intermediate-risk pulmonary embolism. Circulation. 2014 Jan 28;129(4):479-86. doi: 10.1161/CIRCULATIONAHA.113.005544. Epub 2013 Nov 13. PMID 24226805
- [Background] Kuo WT, Banerjee A, Kim PS, DeMarco FJ Jr, Levy JR, Facchini FR, Unver K, Bertini MJ, Sista AK, Hall MJ, Rosenberg JK, De Gregorio MA. Pulmonary Embolism Response to Fragmentation, Embolectomy, and Catheter Thrombolysis (PERFECT): Initial Results From a Prospective Multicenter Registry. Chest. 2015 Sep;148(3):667-673. doi: 10.1378/chest.15-0119. PMID 25856269
- [Background] Piazza G, Hohlfelder B, Jaff MR, Ouriel K, Engelhardt TC, Sterling KM, Jones NJ, Gurley JC, Bhatheja R, Kennedy RJ, Goswami N, Natarajan K, Rundback J, Sadiq IR, Liu SK, Bhalla N, Raja ML, Weinstock BS, Cynamon J, Elmasri FF, Garcia MJ, Kumar M, Ayerdi J, Soukas P, Kuo W, Liu PY, Goldhaber SZ; SEATTLE II Investigators. A Prospective, Single-Arm, Multicenter Trial of Ultrasound-Facilitated, Catheter-Directed, Low-Dose Fibrinolysis for Acute Massive and Submassive Pulmonary Embolism: The SEATTLE II Study. JACC Cardiovasc Interv. 2015 Aug 24;8(10):1382-1392. doi: 10.1016/j.jcin.2015.04.020. PMID 26315743